CLINICAL TRIAL: NCT03656653
Title: Clinical Study of Imagery-based Coping for Cocaine Use Disorder
Brief Title: Imagery-based Coping for Cocaine Use Disorder
Acronym: CIIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: King's College London (Other)
Collaborators: South London and Maudsley NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18?LO/1013
Record Dates: First submitted 2018-08-22; First posted 2018-09-04 (Actual); Last update posted 2019-02-28 (Actual); Status verified 2018-08

CONDITIONS: Cocaine Use Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Future-based recovery-oriented imagery (Experimental): Mental Imagery for Craving Reduction: mental imagery aimed at describing a future without cocaine use
  Interventions: Behavioral: Mental Imagery for Craving Reduction
- Future-based cocaine-aversive imagery (Experimental): Mental Imagery for Craving Reduction: mental imagery aimed at describing a future where cocaine is causing significant distress
  Interventions: Behavioral: Mental Imagery for Craving Reduction
- Past recovery-oriented imagery (Experimental): Mental Imagery for Craving Reduction: mental imagery aimed at describing a past event without cocaine use
  Interventions: Behavioral: Mental Imagery for Craving Reduction
- Past cocaine-aversive imagery (Experimental): Mental Imagery for Craving Reduction: mental imagery aimed at describing a past event where cocaine use has caused significant distress
  Interventions: Behavioral: Mental Imagery for Craving Reduction

INTERVENTIONS:
Behavioral: Mental Imagery for Craving Reduction — a behavioural mental imagery intervention where participants are asked to generate specific mental images to reduce cue-induced craving for cocaine use disorder

SUMMARY:
A pragmatic, 4-week, 4-group, between-subjects, factorial randomised controlled trial conducted at a specialist NHS outpatient addictions clinic and hospital clinical research facility to determine if mental imagery (of past and future positive [recovery oriented] and negative [cocaine aversive] events) can help reduce cue-induced cocaine craving and cocaine use.

DETAILED DESCRIPTION:
Cocaine, a powerful stimulant drug, is used by 2.2% of people aged 16-59 in England and each year about 150.000 people seek help for cocaine use disorder from the NHS or non-governmental organisations (NGO). There are currently no approved medication-assisted treatments or specific psychosocial interventions for CUD. General counselling is offered by the NHS and NGO addiction services, but this is not particularly effective.

The transition from regular cocaine use to cocaine abuse is often marked by intense episodes (binges), which may last several days and are followed by a 'crash' with no or little use. For many people, repeated administration of cocaine over a short duration of time creates vivid episodic memories of euphoria which can inform future craving content. Craving or strong urges are a distinctive feature of CUD and are often reported as involuntary, distressing and uncontrollable.

Research has demonstrated that craving experiences can be voluntarily evoked or elicited by conditioned drug cues in the environment and internal processes such mood or physical sensations. The associations between cues and use are established through classical and instrumental reward-based conditioning and are important for the development and maintenance of CUD. Enhanced attention to cocaine cues develops and remains heightened for at least six months into abstinence.

Craving-related experiences are informed by memories of intense reward, physical sensations and include pro-drug beliefs, appraisals, expectancies and vivid mental imagery. Drug-imagery is often initially pleasurable and affectively charged and can motivate drug-seeking behaviour. If impeded or delayed, drug imagery highlights a deficit and can be experienced as distressing and intrusive. Treatment of intrusive images has been successful in various psychological disorders using imagery rescripting. Imagery rescripting has recently been used in memory-focused cognitive therapy to help reduce cocaine craving. Reducing intrusive image-induced negative affect through positive imagery is important for relieving psychological distress but there is also evidence that aversive imagery may reduce maladaptive approach behaviours.

This will be a pragmatic, 4-week, 2x2, between-subjects, factorial randomised controlled trial. It will be conducted at a specialist NHS outpatient addictions clinic (Lorraine Hewitt House; LHH) operated by South London and Maudsley NHS Foundation trust (SLaM) and at the NIHR Wellcome Trust King's Clinical Research Facility (CRF) at King's College Hospital.

Informed consenting adult participants will be randomised to one of four conditions:

* future-based (prospective) recovery-oriented imagery;
* future-based (prospective) cocaine-aversive imagery;
* past (autobiographical) recovery-oriented imagery; or
* past (autobiographical) cocaine-aversive imagery.

Participants will undergo a craving induction procedure designed to elicit cue-induced craving. In response to elevated craving, participants will be asked to reduce their craving levels using a mental imagery intervention.

Following the procedure in the research facility, participants will be given a digital audio player to take home. This will contain a recording of the imagery condition they are allocated to. Participants will be asked to listen to this recording each day during a 14-day follow-up, and ad libertatem when experiencing cocaine craving. After 14 days participants will be invited for a follow up conducted at the community addictions clinic.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18 years and over; no upper limit);
* English speaking (to a level sufficient to engage with a psychosocial intervention);
* Current diagnosis for primary CUD alone, with concurrent opiate use disorder or while enrolled in opioid agonist therapy *
* Self-reported regular use of crack cocaine;
* Stated motivation to reduce or quit cocaine use;

Exclusion Criteria:

* Current post-traumatic stress disorder (PTCI score >100);
* Suicide attempt in the past 3 months;
* Participants with harmful alcohol consumption (>50 units per week men; >35 units women);
* Cocaine hydrochloride (powder form) users; **
* Non-English Speaking;
* Clinically significant on-going medical problems that might make participation unsafe;
* Uncontrolled Mental Health Disorder;
* Severe neurocognitive impairment (Montreal Cognitive Assessment <17);
* Current enrolment in an addiction treatment related clinical research study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-10-30 (Actual); Primary Completion 2020-01-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Changes in Number of Days abstinent from Cocaine | baseline (Week 0) and at two week-follow up (Week 4)
  The primary outcome measure will be number of days abstinent from cocaine (percentage). A higher percentage indicates a higher number of abstinent days from cocaine.
  This will be expressed as the cumulative distribution function for change (between baseline and follow-up) using a Timeline Follow Back method (calendar prompt).
  Percentage days abstinent is measured for two weeks before the first assessment and two weeks post craving-induction procedure.

SECONDARY OUTCOMES:
Change from baseline in Craving Experience Questionnaire Score (CEQ-12) | baseline (Week 0) and at two week-follow up (Week 4)
  The CEQ-12 is an 12-item, self-report instrument measuring intensity, imagery and intrusiveness dimensions of craving. Each item is rated on a 11-point scale (0-10), ranging from 0-120, where a higher score expresses increased craving.
  The intensity subscale ranges from 0 to 30 where 30 indicates a constant urge to use cocaine.
  The imagery subscale ranges from 0 to 60 where 60 indicates a constant sensory craving experience The intrusiveness subscale ranges from 0 to 30 where 30 indicates constant intrusive thoughts about cocaine
  The CEQ-12 is measured at baseline (craving for past 2 weeks) and at two week-follow up (craving for past two weeks)
  The total craving score will be expressed as cumulative distribution function for change in cocaine craving.
Urine toxicology Screening (UDS) | Assessed at two-week follow up (Week 4)
  By instant result immunoassay device for cocaine metabolite (benzoylecgonine) and morphine (Alere Toxicology).
Imagery Monitoring Diary | Diary assessed at two-week follow up (Week 4)
  A monitoring diary used by participants to indicate use of guided imagery audio and changes in craving levels. Diary will be used daily throughout 14-day follow-up period.
Heart Rate Variability (HRV) | Week 2; 2 hour session
  Real-time HRV data will be acquired through an E4 Empatica (www.empatica.com) wristband placed on the participants' wrist during the craving induction procedure and imagery intervention conducted at the clinical research facility. the HRV is derived from blood volume pulse and will be computed using the mean differences and peak values of the parameters.
Electrodermal Activity (EDA) | Week 2; 2 hour session
  Real-time EDA data will be acquired through an E4 Empatica (www.empatica.com) wristband placed on the participants' wrist during the craving induction procedure and imagery intervention conducted at the clinical research facility. the EDA will be computed using the mean differences and peak values of the parameters.
Temperature | Week 2; 2 hour session
  Real-time EDA data will be acquired through an E4 Empatica (www.empatica.com) wristband placed on the participants' wrist during the craving induction procedure and imagery intervention conducted at the clinical research facility. the EDA will be computed using the mean differences and peak values of the parameters.
Episodic Foresight Score (EFS) | EFS is assessed during the assessment session (Week 1)
  based on the Adapted Autobiographical Interview (AI (Levine et al. 2002; adapted version, Addis, Wong and Schacter (2008)); adapted for this study. The Episodic foresight score (EFS) provides an index of the extent to which participants are personally experiencing an event during mental imagining. This translates into episodic foresight capabilities.
  EFS is derived from transcribed mental image descriptions. Details are segmented and categorised as either internal or external. The number of internal details provided an index of the extent to which participants are personally experiencing the event during mental imagining.
  High score of external details/ Low score of internal detail signify limited episodic foresight whereas a low score of external detail/high score of internal detail signifies good episodic foresight.
Substance Related Imagery Semi Structured Interview (SRI) | Week 1 (Assessment)
  A semi structured interview examining intrusive imagery in substance use. This interview will be used to explore individual craving experiences and help prepare the participant for the imagery intervention.
  Consists of 21 questions exploring imagery in substance use. These are divided into three sections: Exploring Substance Related Images, Link to memories and Negative Valence Imagery.
  Interview consists of a mix of open-ended questions, visual analogue scales and Yes/No questions.
  The interview schedule will be used during the craving experiences interview in the stage 1 assessment.
Predominance of verbal and imagery-based thoughts visual analogue scale (PV-IT) | Week 2 ( x2; Post Craving Induction; Post Imagery Intervention)
  Consists of two rating questions to assess the use of imagery versus verbal thought;
  'How much of the time has your thinking taken the form of verbal thoughts over the past 5 minutes?', 'How much of the time has your thinking taken the form of mental imagery over the past 5 minutes?',
  along with two analogue scales ranging from 'none of the time' to 'all of the time', from 0-9 where 9 indicates all of the time. A higher score indicates frequency of thought in either a visual or verbal modality.
  Scale will be administered post craving induction procedure and post imagery intervention.
The Positive and Negative affect Schedule (PANAS) | Week 2 ( Post Imagery Intervention)
  A self-report questionnaire to measure positive and negative affect. The PANAS consists of 20 different affect-related words. Participants indicate if and to what extent they experience the described feeling at the moment of filling in the questionnaire. The scale ranges from 1-5, where 5 indicates a strong experience of a feeling whereas 1 indicates very slightly or not at all.
  The PANAS provides two scores, one for negative affect and one for positive affect, where higher scores indicate higher levels of negative and positive affect respectively.
  The PANAS will be administered post imagery intervention.
Obsessive Compulsive Drug Use Scale (OCDUS) | Week 1 ( Assessment)
  A self-report questionnaire to measure craving with a focus on the intrusive, obsessive and compulsive characteristics associated to cocaine craving and use.
  The OCDUS has 12 questions rated on a 1-5 Likert Scale and is divided into three subscales: Cocaine Thoughts and Interference (six items), Desire and Control (four items); Resistance to Thoughts and Intention (two items).
  High scores indicate high levels of cocaine thoughts and interference, high levels of desire and low control over cocaine use and low levels of resistance to cocaine thoughts.
  Questionnaire will be administered during Stage 1 assessment.
Patient Health Questionnaire (PHQ-9) | Week 1 (Assessment)
  A self-administered questionnaire to assess depression severity using the DSM-IV depression criteria. The PHQ-9 consists of 9 items rated on a 4 point scale ( 0-3). The PHQ-9 explores the frequency of problems over the last two weeks where 0 is not at all and 3 is nearly every day.
  The total score indicates depression severity as follows: 0-4 none, 5-9 mild, 10-14 moderate, 15-19 moderately severe, 20-27 severe.
  Questionnaire will be administered during Stage 1 assessment.
Generalised Anxiety Disorder Assessment (GAD-7) | Week 1 (Assessment)
  A self-administered questionnaire to assess general anxiety disorder (GAD) using the DSM-IV criteria. The GAD-7 consists of 7 items rated on a 4 point scale ( 0-3). The GAD-7 explores the frequency of problems over the last two weeks where 0 is not at all and 3 is nearly every day.
  The total score (0-21) indicates anxiety severity as follows: : 0-5 mild 6-10 moderate 11-15 moderately severe anxiety ;15-21 severe anxiety.
  Questionnaire will be administered during Stage 1 assessment.

CONTACTS AND LOCATIONS:
Overall Officials: John Marsden, Principal Investigator — King's College London
Locations (1):
- Lorraine Hewitt House, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No